CLINICAL TRIAL: NCT00090571
Title: Research Registry for Juvenile Arthritis
Brief Title: Juvenile Rheumatoid Arthritis Research Registry
Status: Completed | Type: Observational
Sponsor: National Institute of Arthritis and Musculoskeletal and Skin Diseases (NIAMS) (NIH)
Collaborators: Children's Hospital Medical Center, Cincinnati (Other)
Responsible Party: Sponsor
Other Study IDs: NIAMS-102; N01AR42272-8-0-1 (NIH); NIAMS-102;N01-04-03 (Other: NIAMS, NIH)
Record Dates: First submitted 2004-08-27; First posted 2004-08-30 (Estimated); Last update posted 2022-09-28 (Actual); Status verified 2022-09

CONDITIONS: Juvenile Rheumatoid Arthritis
Keywords: JRA ASPs; Genomics
MeSH Terms: conditions — Arthritis, Juvenile

STUDY DESIGN:
Observational Model: Family Based | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — whole blood, serum, Pax gene
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Sib Pairs: Two or more biological siblings affected with JIA.

SUMMARY:
Juvenile rheumatoid arthritis (JRA) is the most common chronic inflammatory disease in children, and may be related to genetics. Having two siblings who both have JRA in one family is rare. The purpose of this registry is to collect patient information and blood samples from qualifying JRA siblings and their families. The goal of the registry is to further understanding of JRA as related to genetics.

DETAILED DESCRIPTION:
JRA is the most common chronic inflammatory pediatric rheumatic disease. JRA may be related to a complex genetic trait. It is rare to have two or more affected siblings, or sibpairs, within one family. The JRA ASP (Affected Sibpair) Registry is a nationwide effort and will collect information and blood samples from JRA sibpairs and their families. Unaffected family members (e.g., mother, father, and unaffected children) are also invited to participate.

Patients and their families may enroll in the registry in one of two ways: patients may contact the registry directly, or they may be referred to the registry through their physician. Once the family has qualified to join the registry, the family will be asked to complete a questionnaire on the medical history of their JRA-affected members. Physicians of the JRA-affected members will be asked to complete questionnaires about their patients' conditions. Family members will also be invited to provide a one-time blood sample. Information collected through the registry will help researchers identify genes involved in JRA susceptibility.

ELIGIBILITY:
Inclusion Criteria for Patients and Their Families:

* At least two members of a family diagnosed with juvenile rheumatoid arthritis (JRA)
* Informed consent from the family indicating willingness to participate in the registry

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: siblings affected with JIA
Sampling Method: Non-Probability Sample
Enrollment: 200 (Actual)
Dates: Start 1994-10; Primary Completion 2009-09 (Actual); Study Completion 2009-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David N. Glass, MD, Principal Investigator — Children's Hospital Medical Center, Cincinnati
Locations (1):
- Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio, United States

REFERENCES:
- [Background] Moroldo MB, Chaudhari M, Shear E, Thompson SD, Glass DN, Giannini EH. Juvenile rheumatoid arthritis affected sibpairs: extent of clinical phenotype concordance. Arthritis Rheum. 2004 Jun;50(6):1928-34. doi: 10.1002/art.20292. PMID 15188369
- [Background] Barnes MG, Aronow BJ, Luyrink LK, Moroldo MB, Pavlidis P, Passo MH, Grom AA, Hirsch R, Giannini EH, Colbert RA, Glass DN, Thompson SD. Gene expression in juvenile arthritis and spondyloarthropathy: pro-angiogenic ELR+ chemokine genes relate to course of arthritis. Rheumatology (Oxford). 2004 Aug;43(8):973-9. doi: 10.1093/rheumatology/keh224. Epub 2004 May 18. PMID 15150433
- [Background] Ogilvie EM, Fife MS, Thompson SD, Twine N, Tsoras M, Moroldo M, Fisher SA, Lewis CM, Prieur AM, Glass DN, Woo P. The -174G allele of the interleukin-6 gene confers susceptibility to systemic arthritis in children: a multicenter study using simplex and multiplex juvenile idiopathic arthritis families. Arthritis Rheum. 2003 Nov;48(11):3202-6. doi: 10.1002/art.11300. PMID 14613283
- [Background] Moroldo MB, Tague BL, Shear ES, Glass DN, Giannini EH. Juvenile rheumatoid arthritis in affected sibpairs. Arthritis Rheum. 1997 Nov;40(11):1962-6. doi: 10.1002/art.1780401107. PMID 9365084
- [Background] Prahalad S, Shear ES, Thompson SD, Giannini EH, Glass DN. Increased prevalence of familial autoimmunity in simplex and multiplex families with juvenile rheumatoid arthritis. Arthritis Rheum. 2002 Jul;46(7):1851-6. doi: 10.1002/art.10370. PMID 12124869
- [Background] Prahalad S, Ryan MH, Shear ES, Thompson SD, Glass DN, Giannini EH. Twins concordant for juvenile rheumatoid arthritis. Arthritis Rheum. 2000 Nov;43(11):2611-2. doi: 10.1002/1529-0131(200011)43:113.0.CO;2-T. No abstract available. PMID 11083290
- [Background] Prahalad S, Ryan MH, Shear ES, Thompson SD, Giannini EH, Glass DN. Juvenile rheumatoid arthritis: linkage to HLA demonstrated by allele sharing in affected sibpairs. Arthritis Rheum. 2000 Oct;43(10):2335-8. doi: 10.1002/1529-0131(200010)43:103.0.CO;2-W. PMID 11037894
- [Background] Hinks A, Ke X, Barton A, Eyre S, Bowes J, Worthington J, Thompson SD, Langefeld CD, Glass DN, Thomson W; UK Rheumatoid Arthritis Genetics Consortium; British Society of Paediatric and Adolescent Rheumatology Study Group. Association of the IL2RA/CD25 gene with juvenile idiopathic arthritis. Arthritis Rheum. 2009 Jan;60(1):251-7. doi: 10.1002/art.24187. PMID 19116909
- [Background] Zeft A, Shear ES, Thompson SD, Glass DN, Prahalad S. Familial autoimmunity: maternal parent-of-origin effect in juvenile idiopathic arthritis. Clin Rheumatol. 2008 Feb;27(2):241-4. doi: 10.1007/s10067-007-0778-8. Epub 2007 Nov 10. PMID 17994193
- [Background] Prahalad S, Bohnsack JF, Whiting A, Clifford B, Jorde LB, Guthery SL, Thompson SD, Glass DN, Bamshad MJ. Lack of association of functional CTLA4 polymorphisms with juvenile idiopathic arthritis. Arthritis Rheum. 2008 Jul;58(7):2147-52. doi: 10.1002/art.23602. PMID 18576317
- [Background] Prahalad S, Bohnsack JF, Jorde LB, Whiting A, Clifford B, Dunn D, Weiss R, Moroldo M, Thompson SD, Glass DN, Bamshad MJ. Association of two functional polymorphisms in the CCR5 gene with juvenile rheumatoid arthritis. Genes Immun. 2006 Sep;7(6):468-75. doi: 10.1038/sj.gene.6364317. Epub 2006 Jun 15. PMID 16775617
- [Background] Phelan JD, Thompson SD. Genomic progress in pediatric arthritis: recent work and future goals. Curr Opin Rheumatol. 2006 Sep;18(5):482-9. doi: 10.1097/01.bor.0000240359.30303.e4. PMID 16896287
- [Background] Phelan JD, Thompson SD, Glass DN. Susceptibility to JRA/JIA: complementing general autoimmune and arthritis traits. Genes Immun. 2006 Jan;7(1):1-10. doi: 10.1038/sj.gene.6364273. PMID 16435022
- [Background] Ferucci ED, Majka DS, Parrish LA, Moroldo MB, Ryan M, Passo M, Thompson SD, Deane KD, Rewers M, Arend WP, Glass DN, Norris JM, Holers VM. Antibodies against cyclic citrullinated peptide are associated with HLA-DR4 in simplex and multiplex polyarticular-onset juvenile rheumatoid arthritis. Arthritis Rheum. 2005 Jan;52(1):239-46. doi: 10.1002/art.20773. PMID 15641089
- [Background] Bukulmez H, Fife M, Tsoras M, Thompson SD, Twine NA, Woo P, Olson JM, Elston RC, Glass DN, Colbert RA. Tapasin gene polymorphism in systemic onset juvenile rheumatoid arthritis: a family-based case-control study. Arthritis Res Ther. 2005;7(2):R285-90. doi: 10.1186/ar1480. Epub 2005 Jan 11. PMID 15743475